CLINICAL TRIAL: NCT03266744
Title: Response Evaluation of Cancer Therapeutics in Metastatic Breast Cancer to the Bone: A Whole Body MRI Study
Acronym: RESPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RD2015-64
Record Dates: First submitted 2017-08-23; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Whole Body MRI; Computerised Tomography; Bone scan
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The reporting radiologist of the WB-MRI will be blinded to the results of the CT. The reporting radiologist of the CT will also be blinded to the results of the WB-MRI. Neither treating clinicians nor patients will be blinded at any point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main study group (Other): Patients will have repeat CT (Computerised Tomography) scans and WB-MRI (Whole Body Magnetic Resonance Imaging) every 12 weeks until disease progression. A baseline bone scan (99mTc-MDP) will be performed.
  At the point of disease progression, a repeat bone scan will be obtained in addition to the CT and WB-MRI.
  Interventions: Diagnostic Test: Computerised Tomography; Diagnostic Test: Whole Body Magnetic Resonance Imaging; Diagnostic Test: Bone scan
- WB-MRI sub-study group (Other): Patients will be given the opportunity to participate in a sub-study of WB-MRI reproducibility. This involves a repeat scan of the Whole Body Magnetic Resonance Imaging (WB-MRI) diffusion-weighted sequences. This will be shorter in duration than the full WB-MRI scan and will take place within one hour of completing the full WB-MRI scan.
  Interventions: Diagnostic Test: Whole Body Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Computerised Tomography
  Arms: Main study group
Diagnostic Test: Whole Body Magnetic Resonance Imaging
Diagnostic Test: Bone scan
  Arms: Main study group

SUMMARY:
This trial is a feasibility study prior to a planned phase III trial. Currently, assessing response to treatment of metastatic breast cancer in the bone is limited by the technical problems associated with CT scans and bone scans. WB-MRI provides theoretical and practical advantages that allow for more detailed analysis of disease response or progression. This may allow for earlier identification of progressive disease and earlier change in treatment.

Participants in the study will have a CT scan, bone scan and WB-MRI at baseline and then repeated CT and WB-MRI scans every 12 weeks (until week 96, and then every 24 weeks) until there is evidence of progressive disease on either of the imaging modalities. In addition to the regular scans on the study, patients will be given the opportunity to participate in a study of how reproducible the findings of WB-MRI scans are. At the point of disease progression, a repeat bone scan is performed and the involvement of the patient in the trial comes to an end.

DETAILED DESCRIPTION:
Patients are eligible for RESPECT if they have bone-only metastatic breast cancer (MBC), as established by standard CT and bone scintigraphy, and are starting a new line of systemic therapy. This can be first line SACT or any subsequent line.

All patients undergo a baseline CT scan (thorax/abdomen/pelvis) and isotope bone scan prior to commencing their new systemic therapy. All CT and bone scans are performed according to standard departmental protocols, with no deviations required. WB-MRI are performed within 2 weeks of study entry. CT scans and WB-MRI are then performed every 12 weeks until week 96, and then every 24 weeks until the patient completes the study. The reporting radiologist who interprets the CT scans is blinded to the images and results of the WB-MRI scan and vice versa.

At study commencement Participants are required to have had a CT scan of the thorax, abdomen and pelvis and a bone scan (bone scintigraphy with technetium-99m-methylene diphosphonate) no more than 4 weeks prior to trial entry to ensure that they have bony-only metastatic disease, as defined using standard imaging. Baseline WB-MRI scans are performed within 2 weeks of entry into the study.

Participants are assessed in clinic and a baseline physical examination is undertaken. Any additional tests required for the initiation of the new SACT are performed at the discretion of the treating clinician and according to local protocols.

During the study CT scans and WB-MRI are performed every 12 weeks until week 96, and then every 24 weeks until disease progression is evident (as defined in the study protocol). Scans are performed within the range of 7 days prior and 7 days after the planned 12 weekly scan interval date.

If there is evidence of equivocal disease progression on WB-MRI only, a repeat WB-MRI is undertaken between 28 and 42 days after the equivocal WB-MRI to confirm or refute the presence of progressive disease. If this confirmed disease progression, then the date of progression is defined as that of the original WB-MRI (i.e. the one performed 4-6 weeks earlier). No repeat CT scans are performed alongside the confirmatory WB-MRI.

Participants are reviewed in outpatient clinic after every imaging time point so that the results of the CT and WB-MRI can be relayed to them by their oncologist and a decision can be made about their ongoing treatment. If more frequent clinic reviews are required then these are not prohibited by the trial protocol. As with the frequency of imaging, the required trial clinic visits change to every 24 weeks after the week 96 visit. During these clinic visits a clinical assessment is made and a full physical examination undertaken. Current anti-cancer drug therapy, including any changes, are documented. Any skeletal related events are also documented. Skeletal related events are defined within the RESPECT study as:

* pathological fracture
* metastatic spinal cord compression
* radiotherapy for bone pain
* surgery to site of bone metastasis Case report forms are completed by the trial administrators at every imaging time point. These are referred to as week 12, week 24, week 36 and so forth.

Patient Imaging Questionnaires are performed at the week 12 and week 36 visits, and are completed by the patients within the radiology department soon after their CT and WB-MRI scans has been performed.

End of study

The end of the study protocol is reached when any of the following occur:

1. Progressive bone and/or visceral disease is demonstrated on CT scan and WB-MRI (as defined in section X).
2. Unequivocal progressive bone and/or visceral disease is demonstrated on WB-MRI alone (as defined in section X).
3. CT and/or WB-MRI findings requiring intervention such as palliative radiotherapy, or a change in systemic therapy.
4. Equivocal evidence of progressive bone and/or visceral disease (not meeting the full criteria for disease progression in section 7.1.3) demonstrated on WB-MRI only, with confirmation of findings on repeat WB-MRI undertaken 4-6 weeks later.
5. Symptomatic skeletal disease or evidence of clinical progression of disease that necessitates a change in systemic therapy.

A repeat nuclear medicine bone scan is undertaken once the participant met one of the end of study criteria above.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of breast cancer
* Single or multiple bone metastases (no extraosseous or non-bony metastatic disease permitted)
* Due to start a new line of either hormone therapy or chemotherapy (use of bisphosphonates / denosumab or targeted agents e.g. trastuzumab in addition to hormone therapy / chemotherapy permitted)
* Aged 18 and over
* Life expectancy of over 6 months
* No current active malignancy other than breast cancer
* Written informed consent must be given according to GCP, and national/local regulations

Exclusion Criteria:

* Radical treatment to sole site of metastatic disease e.g. Cyberknife to solitary bone metastasis
* Absolute contraindication to MRI studies, CT scans or bone scans
* Pregnancy
* Psychological, familial, sociological or geographical conditions that would hamper compliance with the study protocol; such conditions should be discussed with the patient before registration in the trial before patient registration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-04-21 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Disease progression on CT and/or WB-MRI | Up to 96 weeks (from date of consent until the date of first documented progression)
  Description of the metric used to characterize the specific primary outcome measure, if not included in the primary outcome measure title.

SECONDARY OUTCOMES:
Disease progression on CT and/or WB-MRI | Up to 96 weeks (from date of consent until the date of first documented progression)
  Time point(s) at which the measurement is assessed for the specific metric used. The description of the time point(s) of assessment must be specific to the outcome measure and is generally the specific duration of time over which each participant is assessed (not the overall duration of the study).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Andreas Makris, Principal Investigator — East and North Hertfordshire NHS Trust

IPD SHARING:
Plan to Share IPD: Undecided
All patients can agree to their data being used for future research.

REFERENCES:
- [Derived] Kosmin M, Padhani AR, Gogbashian A, Woolf D, Ah-See ML, Ostler P, Sutherland S, Miles D, Noble J, Koh DM, Marshall A, Dunn J, Makris A. Comparison of Whole-Body MRI, CT, and Bone Scintigraphy for Response Evaluation of Cancer Therapeutics in Metastatic Breast Cancer to Bone. Radiology. 2020 Dec;297(3):622-629. doi: 10.1148/radiol.2020192683. Epub 2020 Oct 20. PMID 33078998